CLINICAL TRIAL: NCT00130793
Title: A Double-Blind, Randomized, Controlled, Multicenter Study to Evaluate the Safety, Tolerability and Immunogenicity of a Refrigerator-Stable Formulation of Zoster Vaccine Live (Oka/Merck)
Brief Title: A Study to Evaluate Safety, Tolerability, and Immunogenicity of an Investigational Zoster Vaccine In Subjects With a History of Varicella (Chickenpox)(V211-010)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-010; 2005_035
Record Dates: First submitted 2005-08-11; First posted 2005-08-16 (Estimated); Results first posted 2009-07-03 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- zoster vaccine live (Oka/Merck) refrigerated formulation (Experimental): ZOSTAVAX™ with phosphate-gelatin-sucrose-urea (PGSU) stabilizer (~45,000 plaque-forming units [PFU]), 1 subcutaneous 0.65-mL injection
  Interventions: Biological: Comparator: zoster vaccine live (Oka/Merck) refrigerated formulation
- zoster vaccine live (Oka/Merck) frozen formulation (Active Comparator): ZOSTAVAX™ with phosphate-gelatin-sucrose (PGS) stabilizer (~57,000 PFU), 1 subcutaneous 0.65-mL injection
  Interventions: Biological: Comparator: zoster vaccine live (Oka/Merck) frozen formulation

INTERVENTIONS:
Biological: Comparator: zoster vaccine live (Oka/Merck) refrigerated formulation — 1 dose of 0.65-mL/dose subcutaneous injection of zoster vaccine live (Oka/Merck) refrigerated formulation at Day 1
  Arms: zoster vaccine live (Oka/Merck) refrigerated formulation
Biological: Comparator: zoster vaccine live (Oka/Merck) frozen formulation — 1 dose of 0.65-mL/dose subcutaneous injection of zoster vaccine live (Oka/Meck) frozen formulation at Day 1
  Arms: zoster vaccine live (Oka/Merck) frozen formulation

SUMMARY:
The purpose of this study is to determine whether the refrigerator-stable formulation of an investigational vaccine has a comparable immune response (the body's ability to protect against disease) and safety profile to that of the freezer-stable formulation of the vaccine.

DETAILED DESCRIPTION:
The duration of treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are at least 50 years of age or older with a history of varicella (chicken pox)

Exclusion Criteria:

* Prior history of herpes zoster (shingles)
* Prior receipt of varicella or zoster vaccine
* Immunosuppressed

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2005-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Gilderman LI, Lawless JF, Nolen TM, Sterling T, Rutledge RZ, Fernsler DA, Azrolan N, Sutradhar SC, Wang WW, Chan IS, Schlienger K, Schodel F, Silber JL; Zostavax Protocol 010 Study Group. A double-blind, randomized, controlled, multicenter safety and immunogenicity study of a refrigerator-stable formulation of Zostavax. Clin Vaccine Immunol. 2008 Feb;15(2):314-9. doi: 10.1128/CVI.00310-07. Epub 2007 Dec 12. PMID 18077611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 14 sites in the United States.
  First patient randomized: 08Aug2005; Last patient last visit: 28Nov2005
Groups:
- ZOSTAVAX™ With PGSU: ZOSTAVAX™ with phosphate-gelatin-sucrose-urea (PGSU) stabilizer (~45,000 plaque-forming units [PFU]), 1 subcutaneous 0.65-mL injection
- ZOSTAVAX™ With PGS: ZOSTAVAX™ with phosphate-gelatin-sucrose (PGS) stabilizer (~57,000 PFU), 1 subcutaneous 0.65-mL injection
Period: Overall Study
Arm/Group | ZOSTAVAX™ With PGSU | ZOSTAVAX™ With PGS
Started | 183 | 185
Vaccinated | 182 (One subject was allocated but not vaccinated.) | 185
Completed | 180 (Subject received vaccine, completed blood draws, returned vaccination report card (VRC) at Week 4) | 181 (Subject received vaccine, completed blood draws, returned VRC at Week 4)
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrew consent | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX™ With PGSU | ZOSTAVAX™ With PGS | Total
Number analyzed (Participants) | 182 | 185 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.25) | 63.2 (8.44) | 63.35 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 106 | 203
  Male | 85 | 79 | 164
Race/Ethnicity [Number; unit: participants]
  Asian | 6 | 6 | 12
  Asiatic | 1 | 4 | 5
  Black | 19 | 15 | 34
  Hispanic American | 30 | 34 | 64
  Indian | 1 | 0 | 1
  Native American | 1 | 0 | 1
  White | 124 | 126 | 250

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Varicella-zoster Virus (VZV) Antibody Responses at 4 Weeks Postvaccination
Description: The GMT of the VZV-specific antibody responses as measured by gpELISA (glycoprotein enzyme-linked immunosorbent assay) at 4 weeks postvaccination in subjects who received ZOSTAVAX™ with PGSU and in subjects who received ZOSTAVAX™ with PGS.
Time Frame: 4 weeks
Population: The primary immunogenicity analyses were based on the per-protocol population defined as subjects who had valid results from samples obtained within the prespecified day ranges at Day 1 or at Week 4 postvaccination, and who did not meet any of the protocol violations prespecified in the statistical analysis plan (SAP)
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | ZOSTAVAX™ With PGSU | ZOSTAVAX™ With PGS
Number analyzed (Participants) | 176 | 178
gpELISA units/mL | 717.5 [607.3 to 847.7] | 844.9 [704.4 to 1013.6]

2. Secondary Outcome: Vaccine-Related Serious Adverse Experiences (SAEs) for 28 Days Postvaccination
Description: Vaccine-related (as assessed by an investigator who is a qualified physician according to his/her best clinical judgment) serious adverse experiences are any AEs occurring at any dose that; Results in death; or Is life threatening; or Results in a persistent or significant disability/incapacity; or Results in or prolongs an existing inpatient hospitalization; or Is a congenital anomaly/birth defect; or Is a cancer; or Is an overdose
Time Frame: 4 weeks
Population: All vaccinated subjects with safety follow-up are included.
Measure: Number; unit: Participants
Arm/Group | ZOSTAVAX™ With PGSU | ZOSTAVAX™ With PGS
Number analyzed (Participants) | 180 | 183
Participants
  With vaccine related SAEs | 0 | 0
  Without vaccine related SAEs | 180 | 183

3. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titers From Prevaccination to 4 Weeks Postvaccination
Description: GMFR of the VZV antibody response from prevaccination to Week 4 postvaccination
Time Frame: From prevaccination (baseline) to 4 weeks postvaccination
Population: The primary immunogenicity analyses were based on the per-protocol population defined as subjects who had valid results from samples obtained within the prespecified day ranges at Day 1 or at Week 4 postvaccination, and who did not meet any of the protocol violations prespecified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Groups:
- ZOSTAVAX™With PGSU: ZOSTAVAX™with phosphate-gelatin-sucrose-urea (PGSU) stabilizer (~45,000 plaque-forming units [PFU]), 1 subcutaneous 0.65-mL injection
Arm/Group | ZOSTAVAX™With PGSU | ZOSTAVAX™ With PGS
Number analyzed (Participants) | 174 | 177
gpELISA units/mL | 2.6 [2.2 to 3.0] | 2.9 [2.4 to 3.4]

ADVERSE EVENTS:
Time Frame: Through 28 days post-vaccination.
Description: The AE presentation includes participants who were vaccinated and had safety follow-up.
Arm/Group | ZOSTAVAX™ With PGSU | ZOSTAVAX™ With PGS
Serious Adverse Events (participants affected / at risk) | 1/180 | 0/183
Other Adverse Events (participants affected / at risk) | 63/180 | 84/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZOSTAVAX™ With PGSU (N=180) | ZOSTAVAX™ With PGS (N=183)
Gastroenteritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZOSTAVAX™ With PGSU (N=180) | ZOSTAVAX™ With PGS (N=183)
Injection site erythema (General disorders) | 52 | 65
Injection site pain (General disorders) | 48 | 70
Injection site pruritus (General disorders) | 13 | 16
Injection site swelling (General disorders) | 44 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.